CLINICAL TRIAL: NCT05014438
Title: A Phase 2, Randomized, Double-blinded, Placebo-controlled, 5 Parallel-group Study of BMS-986166 or Branebrutinib for the Treatment of Patients With Moderate to Severe Atopic Dermatitis
Brief Title: A Study of BMS-986166 or Branebrutinib for the Treatment of Participants With Atopic Dermatitis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: IM018-005; 2020-004767-77 (EudraCT Number); U1111-1259-1220 (Registry Identifier: WHO)
Record Dates: First submitted 2021-07-29; First posted 2021-08-20 (Actual); Results first posted 2023-10-18 (Actual); Last update posted 2023-10-18 (Actual); Status verified 2023-09

CONDITIONS: Dermatitis, Atopic
Keywords: Atopic Dermatitis; BMS-986166; BMS-986195; Branebrutinib
MeSH Terms: conditions — Dermatitis, Atopic | interventions — BMS-986166; branebrutinib

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- Placebo (Placebo Comparator)
  Interventions: Other: Placebo
- Treatment BMS-986166 Dose 1 (Experimental)
  Interventions: Drug: BMS-986166
- Treatment BMS-986166 Dose 2 (Experimental)
  Interventions: Drug: BMS-986166
- Treatment BMS-986166 Dose 3 (Experimental)
  Interventions: Drug: BMS-986166
- Treatment Branebrutinib (Experimental)
  Interventions: Drug: Branebrutinib

INTERVENTIONS:
Drug: BMS-986166 — Specified dose on specified days
  Arms: Treatment BMS-986166 Dose 1; Treatment BMS-986166 Dose 2; Treatment BMS-986166 Dose 3
Drug: Branebrutinib — Specified dose on specified days
  Other Names: BMS-986195
  Arms: Treatment Branebrutinib
Other: Placebo — Specified dose on specified days
  Arms: Placebo

SUMMARY:
The purpose of this study is to evaluate the efficacy, safety, and tolerability of BMS-986166 and of branebrutinib, each versus placebo, for the treatment of participants with moderate to severe atopic dermatitis.

ELIGIBILITY:
Inclusion Criteria:

* Chronic atopic dermatitis (AD) diagnosed according to the Eichenfield modification of Hanifin's and Rajka's (E-HR) criteria at Screening
* Disease duration of at least 24 months since diagnosis by any criteria
* Documented history of inadequate control of AD by a stable regimen (≥ 4 weeks) of topical corticosteroids, calcineurin inhibitors or biologics, within 6 months of randomization, or inappropriateness of therapy due to side effects or safety risks leading to prior discontinuation
* Application of fixed doses of an additive-free, basic bland emollient twice-daily for ≥ 7 days before baseline visit and for the duration of the study

Exclusion Criteria:

* Any major illness/condition or evidence of an unstable clinical condition or local active infection/infectious illness that, in the investigator's judgment, will substantially increase the risk to the participant if he or she participates in the study or interfere with the interpretation of study results
* Clinically relevant cardiovascular conditions or pulmonary conditions
* High likelihood - based on participant history, and investigator judgement - of requiring rescue therapy in < 4 weeks prior to randomization
* Evidence of acute flare between the Screening and Baseline/ Randomization
* Skin lesion(s) and/or pruritus due to conditions other than AD that would interfere with the study specified assessments

Other protocol-defined inclusion/exclusion criteria apply

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2021-08-17 (Actual); Primary Completion 2022-08-22 (Actual); Study Completion 2022-08-22 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (42):
- United States (17):
  - Local Institution - 0091, Fremont, California
  - Local Institution - 0112, Brandon, Florida
  - Local Institution - 0061, Coral Gables, Florida
  - Local Institution - 0110, Margate, Florida
  - Local Institution - 0006, Miami Lakes, Florida
  - Local Institution, Tampa, Florida
  - Local Institution - 0008, Skokie, Illinois
  - Local Institution - 0081, Indianapolis, Indiana
  - Local Institution - 0083, Louisville, Kentucky
  - Dermatology and Skin Cancer Specialists, LLC, Rockville, Maryland
  - Local Institution - 0051, Saint Joseph, Missouri
  - Local Institution, New York, New York
  - Local Institution - 0078, Philadelphia, Pennsylvania
  - Local Institution - 0094, Pittsburgh, Pennsylvania
  - The University of Texas Health Science Center at Houston, Bellaire, Texas
  - Local Institution, San Antonio, Texas
  - Local Institution - 0003, Morgantown, West Virginia
- Australia (4):
  - Premier Dermatology, Kogarah, New South Wales
  - Holdsworth House Medical Practice, Sydney, New South Wales
  - Westmead Hospital-Dermatology, Westmead, New South Wales
  - Sinclair Dermatology, East Melbourne, Victoria
- Local Institution, Linz, Austria
- Canada (3):
  - Local Institution, Markham, Ontario
  - York Dermatology Clinic and Research Centre, Richmond Hill, Ontario
  - SIMa Recherche, Verdun, Quebec
- Germany (10):
  - Charité Universitaetsmedizin Berlin - Campus Mitte, Berlin
  - Local Institution, Berlin
  - Local Institution - 0034, Bochum
  - Universitätsklinikum Bonn-Studienzentrum Dermatologie, Bonn
  - SRH Wald-Klinikum Gera-Zentrum für klinische Studien, Gera
  - Local Institution, Hanover
  - Universitatsklinikum Schleswig-Holstein, Kiel
  - Local Institution, Munich
  - KliFOs - Klinische Forschung Osnabrück, Osnabrück
  - Private Practice - Dr. Ralph von Kiedrowski, Selters
- Poland (3):
  - Royalderm Agnieszka Nawrocka, Warsaw, Masovian Voivodeship
  - NZOZ Centrum Medyczne KERmed, Bydgoszcz
  - ETYKA Osrodek Badan Klinicznych, Olsztyn
- Spain (4):
  - Local Institution - 0130, Córdoba, Andalusia
  - Hospital General Universitario de Alicante-Dermatology, Alicante
  - Hospital Universitario de Gran Canaria Doctor Negrín-Dermatología, Las
  - Hospital Universitario La Paz-UCICEC/DERMA, Madrid

REFERENCES:
- See also: BMS Clinical Trial Information — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html
- See also: BMS Clinical Trial Patient Recruiting — http://www.BMSStudyConnect.com

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 17 participants randomized and treated
Groups:
- Placebo: Placebo
- Treatment 1: BMS-986166 0.25mg POQD
- Treatment 2: BMS-986166 0.5mg POQD
- Treatment 3: BMS-986166 0.75mg POQD
- Treatment 4: Branebrutinib 9mg POQD
Period: Overall Study
Arm/Group | Placebo | Treatment 1 | Treatment 2 | Treatment 3 | Treatment 4
Started | 4 | 3 | 4 | 3 | 3
Completed | 3 | 3 | 3 | 1 | 3
Not Completed | 1 | 0 | 1 | 2 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Treatment 1 | Treatment 2 | Treatment 3 | Treatment 4 | Total
Number analyzed (Participants) | 4 | 3 | 4 | 3 | 3 | 17
Age, Continuous [Mean (Standard Deviation); unit: Years] | 30.5 (11.3) | 36.0 (6.2) | 29.5 (14.6) | 46.7 (8.3) | 36.7 (17.8) | 35.2 (12.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 1 | 3 | 2 | 2 | 11
  Male | 1 | 2 | 1 | 1 | 1 | 6
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 0 | 0 | 1 | 1 | 4
  Not Hispanic or Latino | 2 | 3 | 3 | 2 | 2 | 12
  Unknown or Not Reported | 0 | 0 | 1 | 0 | 0 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 1 | 0 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 1 | 0 | 0 | 1
  White | 3 | 3 | 2 | 3 | 3 | 14
  More than one race | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 1 | 0 | 0 | 0 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Mean Percentage Change From Baseline in EASI Score at Week 16
Description: The Eczema Area and Severity Index (EASI) is a validated, composite scoring system assessed by the investigator based on the extent of each of the 4 body regions (head and neck, upper limbs, lower limbs, and trunk) affected with AD and the intensity of each of 4 key signs of AD (erythema, induration/papulation, excoriation, and lichenification) and is based on a 4-point scale of 0 (absent), 1 (mild), 2 (moderate), and 3 (severe). For each of the 4 body regions, the mean intensity of inflamed lesions for each of the 4 signs is recorded. Xerosis, scaling, urticaria, or post-inflammatory pigmentation changes are not included. The total EASI score ranges from 0 to 72.
  The lower the score the better.
Time Frame: From baseline and 16 weeks
Population: mITT population with evaluable EASI score at baseline and week 16. mITT: Modified Intent-To-Treat (All participants who are randomized and received at least one dose of study treatment)
Measure: Mean (Standard Deviation); unit: Percentage change
Arm/Group | Placebo | Treatment 1 | Treatment 2 | Treatment 3 | Treatment 4
Number analyzed (Participants) | 1 | 0 | 0 | 0 | 1
Percentage change | -83.1 (NA) — Insufficient number of participants analyzed to calculate SD |  |  |  | -92.3 (NA) — Insufficient number of participants analyzed to calculate SD

2. Secondary Outcome: Percentage of Participants Exhibiting a Validated Investigator Global Assessment for Atopic Dermatitis (vIGA-AD) Score of 0 (Cleared) or 1 (Almost Cleared) AND a ≥ 2 Point Reduction From Baseline at Week 16
Description: The vIGA-AD is a static 5-point assessment intended to assess the global severities of key acute clinical signs of AD, including erythema, induration/papulation, and oozing/crusting (lichenification excluded).
  The rating of cleared (0), almost cleared (1), mild (2), moderate (3), and severe (4) will be assessed.
Time Frame: From baseline and 16 weeks
Population: mITT population with evaluable vIGA-AD at baseline. mITT: Modified Intent-To-Treat (All participants who are randomized and received at least one dose of study treatment)
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Placebo | Treatment 1 | Treatment 2 | Treatment 3 | Treatment 4
Number analyzed (Participants) | 4 | 3 | 4 | 3 | 3
Percentage of participants | 0 [0.0 to 60.2] | 0 [0.0 to 70.8] | 0 [0.0 to 60.2] | 0 [0.0 to 70.8] | 0 [0.0 to 70.8]

3. Secondary Outcome: Percentage of Participants Exhibiting a ≥ 50% (EASI-50) Reduction From Baseline in EASI Score at Week 16
Description: as for outcome 1
Time Frame: From baseline and 16 weeks
Population: mITTpopulationIntent-To-Treat (All participants who are randomized and received at least one dose of study treatment)
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Placebo | Treatment 1 | Treatment 2 | Treatment 3 | Treatment 4
Number analyzed (Participants) | 4 | 3 | 4 | 3 | 3
Percentage of participants | 25 [0.6 to 80.6] | 0 [0.0 to 70.8] | 0 [0.0 to 60.2] | 0 [0.0 to 70.8] | 33.3 [0.8 to 90.6]

4. Secondary Outcome: Percentage of Participants Exhibiting a ≥ 4-point Improvement From Baseline in Pruritus NRS at Week 16
Description: Participants will complete a daily diary recording the intensity of their pruritus they experienced during the preceding 24 hours. The intensity of pruritus will be assessed using a validated 11-point NRS, ranging from 0 ("no itching") to 10 ("the worst itching imaginable").
  The lower the score the better.
Time Frame: From baseline and 16 weeks
Population: mITT population with evaluable baseline pruritis NRS greater than or equal to 4. mITT: Modified Intent-To-Treat (All participants who are randomized and received at least one dose of study treatment)
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Placebo | Treatment 1 | Treatment 2 | Treatment 3 | Treatment 4
Number analyzed (Participants) | 4 | 3 | 2 | 2 | 2
Percentage of participants | 25.0 [0.6 to 80.6] | 0 [0.0 to 70.8] | 0 [0.0 to 84.2] | 50 [1.3 to 98.7] | 50 [1.3 to 98.7]

5. Secondary Outcome: Mean Percentage Change From Baseline in Pruritus NRS Score at Week 16
Description: Participants will complete a daily diary recording the intensity of their pruritus and the average quality of sleep they experienced during the preceding 24 hours. The intensity of pruritus will be assessed using a validated 11-point NRS, ranging from 0 ("no itching") to 10 ("the worst itching imaginable"). The quality of sleep will be assessed using a validated 11-point NRS ranging from 0 ("the best possible sleep") to 10 ("the worst possible sleep).
  The lower the score the better.
Time Frame: From baseline and 16 weeks
Population: mITT population with evaluable Pruritus NRS at baseline and week 16. mITT: Modified Intent-To-Treat (All participants who are randomized and received at least one dose of study treatment)
Measure: Mean (Standard Deviation); unit: Percentage change
Arm/Group | Placebo | Treatment 1 | Treatment 2 | Treatment 3 | Treatment 4
Number analyzed (Participants) | 1 | 0 | 0 | 1 | 1
Percentage change | -89.6 (NA) — Too few participants to calculate SD |  |  | -100 (NA) — Too few participants to calculate SD | -86.8 (NA) — Too few participants to calculate SD

6. Secondary Outcome: Mean Change From Baseline in Percentage of Affected BSA at Week 16
Description: A widely used method of measuring Body Surface Area (BSA) involvement by AD, is the rule of nines in which for each section of the body (the possible highest score for each region is: head and neck [9%], anterior trunk [18%], back [18%], upper limbs [18%], lower limbs [36%], genitals [1%]) and will be reported as a percentage of all major body sections combined.
Time Frame: From baseline and 16 weeks
Population: mITT population with evaluable baseline and week 16 BSA measurement. mITT: Modified Intent-To-Treat (All participants who are randomized and received at least one dose of study treatment)
Measure: Mean (Standard Deviation); unit: Percentage change
Arm/Group | Placebo | Treatment 1 | Treatment 2 | Treatment 3 | Treatment 4
Number analyzed (Participants) | 1 | 0 | 0 | 0 | 1
Percentage change | -17.00 (NA) — Too few participants to calculate SD |  |  |  | -12.10 (NA) — Too few participants to calculate SD

7. Secondary Outcome: Number of Participants With Mild Moderate or Severe AEs
Description: An Adverse Event (AE) is defined as any new untoward medical occurrence or worsening of a pre-existing medical condition in a clinical investigation participant administered study treatment that does not necessarily have a causal relationship with this treatment.
  Mild: An event that is easily tolerated by the participant, causing minimal discomfort and not interfering with everyday activities.
  Moderate: An event that causes sufficient discomfort and interferes with normal everyday activities.
  Severe: An event that prevents normal everyday activities. An AE that is assessed as severe should not be confused with an SAE. Severe is a category utilized for rating the intensity of an event, and both AEs and SAEs can be assessed as severe.
Time Frame: From initial treatment to 30 days post discontinuation, approximately 29 weeks
Population: Safety Population
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Treatment 1 | Treatment 2 | Treatment 3 | Treatment 4
Number analyzed (Participants) | 4 | 3 | 4 | 3 | 3
Participants
  Mild | 1 | 2 | 1 | 1 | 1
  Moderate | 1 | 3 | 1 | 1 | 0
  Severe | 0 | 0 | 0 | 0 | 0

8. Secondary Outcome: Number of Participants With Mild Moderate or Severe SAEs
Description: A Serious Adverse Event (SAE) is defined as any untoward medical occurrence that, at any dose:
  * Results in death
  * is life threatening
  * Requires inpatient hospitalization or causes prolongation of existing hospitalization
  * Results in persistent or significant disability
  * Is a congenital anomaly/birth defect.
  * Is an important medical event
Time Frame: From initial treatment to 30 days post discontinuation, approximately 29 weeks
Population: Safety Population
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Treatment 1 | Treatment 2 | Treatment 3 | Treatment 4
Number analyzed (Participants) | 4 | 3 | 4 | 3 | 3
Participants
  Mild | 0 | 0 | 0 | 0 | 0
  Moderate | 0 | 1 | 0 | 0 | 0
  Severe | 0 | 0 | 0 | 0 | 0

9. Secondary Outcome: Number of Participants With Clinically Relevant ECG Abnormalities
Description: 12 Lead Electrocardiogram (ECG). The participant will remain supine for 5 to 10 minutes prior to the ECG and must have lab work done after the tracing so that the ECG results remain as accurate as possible.
Time Frame: Week 24 after initial treatment
Population: Safety Population
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Treatment 1 | Treatment 2 | Treatment 3 | Treatment 4
Number analyzed (Participants) | 4 | 3 | 4 | 3 | 3
Participants | 0 | 0 | 0 | 0 | 0

10. Secondary Outcome: Number of Participants With Clinically Relevant OCT Abnormalities
Description: Optical coherence tomography (OCT) is a non-invasive imaging test. It uses light waves to take cross-section pictures of your retina. Diagnosis is made by an ophthalmologist.
Time Frame: Week 24 after initial treatment
Population: Safety population
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Treatment 1 | Treatment 2 | Treatment 3 | Treatment 4
Number analyzed (Participants) | 4 | 3 | 4 | 3 | 3
Participants | 0 | 0 | 1 | 0 | 0

11. Secondary Outcome: Number of Participants With Clinically Relevant PFT Abnormalities
Description: Pulmonary function tests (PFT) include: forced expiratory volume (FEV1), percent predicted FEV1, forced vital capacity (FVC), percent predicted FVC, and Diffusion capacity of carbon monoxide (DLCO).
Time Frame: Week 24 after initial treatment
Population: Safety Population
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Treatment 1 | Treatment 2 | Treatment 3 | Treatment 4
Number analyzed (Participants) | 4 | 3 | 4 | 3 | 3
Participants | 0 | 0 | 0 | 0 | 0

12. Secondary Outcome: Number of Participants With Clinically Meaningful Changes in Vital Signs
Description: The following vital signs will be assessed: systolic blood pressure, diastolic blood pressure, heart rate, respiratory rate and body temperature.
Time Frame: Week 24 after initial treatment
Population: Safety Population
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Treatment 1 | Treatment 2 | Treatment 3 | Treatment 4
Number analyzed (Participants) | 4 | 3 | 4 | 3 | 3
Participants
  Respiratory Rate | 2 | 1 | 2 | 3 | 3
  Heart Rate | 0 | 0 | 0 | 0 | 0
  Diastolic Blood Pressure | 0 | 0 | 0 | 0 | 0
  Systolic Blood Pressure | 0 | 0 | 0 | 0 | 0
  Body Temperature | 0 | 0 | 0 | 0 | 0

13. Secondary Outcome: Number of Participants With Clinically Relevant Changes in LFTs
Description: Liver Function Tests (LFTs) will include the following measurements:
  * ALT OR AST > 3 X ULN
  * ALT OR AST > 5 X ULN
  * ALT OR AST > 8 X ULN
  * TOTAL BILIRUBIN > 2 X ULN
  * ALT OR AST > 3 X ULN AND (TOTAL BILIRUBIN > 2 X ULN OR INR >1.5)
  AST = aspartate aminotransferase ALT = alanine aminotransferase ULN = Upper limit number INR = International Normalized Ratio
Time Frame: Week 24 after initial treatment
Population: Safety Population
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Treatment 1 | Treatment 2 | Treatment 3 | Treatment 4
Number analyzed (Participants) | 4 | 3 | 4 | 3 | 3
Participants
  ALT OR AST > 3 X ULN | 0 | 0 | 0 | 0 | 0
  ALT OR AST > 5 X ULN | 0 | 0 | 0 | 0 | 0
  ALT OR AST > 8 X ULN | 0 | 0 | 0 | 0 | 0
  TOTAL BILIRUBIN > 2 X ULN | 0 | 0 | 0 | 0 | 0
  ALT OR AST > 3 X ULN AND (TOTAL BILIRUBIN > 2 X ULN OR INR >1.5) | 0 | 0 | 0 | 0 | 0
  ALT OR AST > 5 X ULN WITH CONFIRMATION, WITHIN 2 WEEKS | 0 | 0 | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: Adverse Events and Serious Adverse Events: (From first dose to last dose + 8 weeks follow up): Approximately 29 Weeks All-Cause mortality (From randomization to end of study): Approximately 29 Weeks
Description: The number at Risk for All-Cause Mortality represents all Randomized Participants. The number at Risk for Serious Adverse Events and Other (Not Including Serious) Adverse Events represents all participants that received at least 1 dose of study medication
Arm/Group | Placebo | Treatment 1 | Treatment 2 | Treatment 3 | Treatment 4
All-Cause Mortality (participants affected / at risk) | 0/4 | 0/3 | 0/4 | 0/3 | 0/3
Serious Adverse Events (participants affected / at risk) | 0/4 | 1/3 | 0/4 | 0/3 | 0/3
Other Adverse Events (participants affected / at risk) | 2/4 | 3/3 | 2/4 | 1/3 | 1/3
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=4) | Treatment 1 (N=3) | Treatment 2 (N=4) | Treatment 3 (N=3) | Treatment 4 (N=3)
Eczema herpeticum (Infections and infestations) | 0 | 1 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=4) | Treatment 1 (N=3) | Treatment 2 (N=4) | Treatment 3 (N=3) | Treatment 4 (N=3)
Lymphadenopathy (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0 | 0
Macular degeneration (Eye disorders) | 0 | 0 | 1 | 0 | 0
Visual impairment (Eye disorders) | 0 | 1 | 0 | 0 | 0
Abdominal pain upper (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0
Nodule (General disorders) | 0 | 1 | 0 | 0 | 0
Pyrexia (General disorders) | 0 | 1 | 0 | 0 | 0
Furuncle (Infections and infestations) | 0 | 1 | 0 | 0 | 0
Nasopharyngitis (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Skin bacterial infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 0 | 1 | 0 | 0 | 0
Diabetes mellitus inadequate control (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1
Hyperuricaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0
Depressed mood (Psychiatric disorders) | 0 | 1 | 0 | 0 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0
Dermatitis atopic (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0
Skin mass (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-06-30): https://cdn.clinicaltrials.gov/large-docs/38/NCT05014438/Prot_SAP_000.pdf